CLINICAL TRIAL: NCT03730337
Title: Open-label, Uncontrolled, Dose-escalation Study of ONO-7475 Given as Monotherapy and Combinations With ONO-4538 in Patients With Advanced or Metastatic Solid Tumors
Brief Title: Phase 1 Study of ONO-7475 With and Without ONO-4538 in Subjects Advanced or Metastatic Solid Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Ono Pharmaceutical Co. Ltd (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ONO-7475-02 / ONO-4538-74
Record Dates: First submitted 2018-10-30; First posted 2018-11-05 (Actual); Last update posted 2023-10-04 (Actual); Status verified 2023-09

CONDITIONS: Advanced or Metastatic Solid Tumors
MeSH Terms: interventions — Nivolumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ONO-7475 monotherapy (Experimental)
  Interventions: Drug: ONO-7475
- ONO-7475 in combination with ONO-4538 (Experimental)
  Interventions: Drug: ONO-7475 + ONO-4538

INTERVENTIONS:
Drug: ONO-7475 — ONO-7475 specified dose on specified days
  Arms: ONO-7475 monotherapy
Drug: ONO-7475 + ONO-4538 — ONO-7475+ONO-4538 specified dose on specified days
  Arms: ONO-7475 in combination with ONO-4538

SUMMARY:
To evaluate the tolerability and safety of ONO-7475 monotherapy and combinations with ONO-4538 in patients with advanced or metastatic solid tumors

ELIGIBILITY:
Inclusion Criteria:

* Patients with histologically or cytologically confirmed advanced or metastatic solid tumors
* ECOG Performance Status 0～1
* Patients with life expectancy of at least 3 months

Exclusion Criteria:

* Patients with history of severe allergy
* Patients with multiple cancers

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2018-10-17 (Actual); Primary Completion 2021-06-28 (Actual); Study Completion 2022-11-22 (Actual)

PRIMARY OUTCOMES:
Number of paticipants with dose-limiting toxicities during the DLT evaluation period | 28 days
Incidence and severity of adverse events as assessed by CTCAE v4.0 to determine the tolerability and safety | Through study completion, an average of 1 year

SECONDARY OUTCOMES:
Pharmacokinetics (Cmax) | Through study completion
  Assessment of the maximum plasma concentration of ONO-7475 both alone and in combination with ONO-4538
Pharmacokinetics (Tmax) | Through study completion
  Assessment of the time to reach maximum observed plasma concentration of ONO-7475 both alone and in combination with ONO-4538
Pharmacokinetics (AUC) | Through study completion
  Assessment of the plasma area under the curve of ONO-7475 both alone and in combination with ONO-4538

CONTACTS AND LOCATIONS:
Overall Officials: Project Leader, Study Director — Ono Pharmaceutical Co. Ltd
Locations (1):
- Tokyo Clinical Site, Tokyo, Japan

REFERENCES:
- [Derived] Zhao X, Li Y, Yang S, Chen Y, Wu K, Geng J, Liu P, Wang Z, Dai H, Wang C. Orderly Regulation of Macrophages and Fibroblasts by Axl in Bleomycin-Induced Pulmonary Fibrosis in Mice. J Cell Mol Med. 2025 Jan;29(1):e70321. doi: 10.1111/jcmm.70321. PMID 39779468